CLINICAL TRIAL: NCT03165032
Title: Right Ventricular Function During Exercise in Highlanders With Pulmonary Hypertension Compared to Highlanders Without Pulmonary Hypertension and Lowlanders
Brief Title: Right Ventricular Function During Exercise in Highlanders/Lowlanders
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Principal Investigator, Silvia Ulrich Somaini, Prof. Dr., University of Zurich
Other Study IDs: 01-8/433B
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: exercise; echocardiography; right ventricular function; pulmonary hypertension; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Motor Activity; Hypertension, Pulmonary; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High altitude pulmonary hypertension: Highlanders with high altitude pulmonary hypertension living above 2500 m.
- High altitude control: Healthy highlanders living above 2500 m.
- Low altitude control: Healthy lowlanders living below 1000 m.

SUMMARY:
The purpose of the current study is to evaluate the right ventricular function during graded cycling on an ergometer by transthoracic echocardiography in Kyrgyz highlanders with high altitude pulmonary hypertension (HAPH) by performing a cross-sectional case-control study.

ELIGIBILITY:
Inclusion Criteria:

* high altitude pulmonary hypertension confirmed by clinical presentation and mean pulmonary artery pressure >30 mmHg measured by echocardiography at altitude of residence.
* healthy subjects (high altitude controls)
* Both genders
* Age >16 y
* Kyrgyz ethnicity
* born, raised and currently living at >2500 m
* healthy subjects currently living at <1000 m (low altitude controls)

Exclusion Criteria:

* Pulmonary hypertension from other causes, in particular from left ventricular failure as judged clinically and by echocardiography
* Excessive erythrocytosis
* Other coexistent disorders that may interfere with the cardio-respiratory system and sleep
* Regular use of medication that affects control of breathing
* Heavy smoking

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Highlanders with high altitude pumonary hypertension living at an altitude of 2500-4000 m; healthy highlanders living at an altitude of 2500-4000 m; healthy lowlanders living at an altitude of <1000 m.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
pulmonary artery pressure (PAP) during exercise | Day 2
  Difference in change of tricuspid pressure gradient during exercise between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography during graded cycling on an ergometer

SECONDARY OUTCOMES:
cardiac output (CO) during exercise | Day 2
  Difference in change of cardiac output during exercise between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography during graded cycling on an ergometer
PAP/CO slope during exercise | Day 2
  Difference in change of PAP/CO slope during exercise between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography during graded cycling on an ergometer
Oxygen saturation | Day 2
  Difference in change of oxygen saturation during exercise between highlanders with pulmonary hypertension, healthy highlanders and healthy lowlanders, measured by transthoracic echocardiography during graded cycling on an ergometer

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided